CLINICAL TRIAL: NCT02739087
Title: Radiation-Free Heart Catheterization Using MRI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joshua Kanter (Other)
Responsible Party: Sponsor-Investigator, Joshua Kanter, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3860; Internal Bridge funding (Other: Children's Research Institute, Children's National)
Record Dates: First submitted 2016-02-17; First posted 2016-04-14 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Aortic Coarctation; Cardiomyopathy; Atrial Septal Defect; Aortic Stenosis; Post Heart Transplant Catheter Procedure; Patent Ductus Arteriosus
Keywords: radiation free cardiac catheterization
MeSH Terms: conditions — Aortic Coarctation; Cardiomyopathies; Heart Septal Defects, Atrial; Aortic Valve Stenosis; Ductus Arteriosus, Patent | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI guided cardiac catheterization (Experimental): Magnetic resonance imaging will be used to guide cardiac catheterization procedures.
  Interventions: Procedure: MRI guided cardiac catheterization; Device: Magnetic resonance imaging

INTERVENTIONS:
Procedure: MRI guided cardiac catheterization — Magnetic resonance imaging will be used to guide cardiac catheterization procedures whenever possible to avoid or minimize x-ray radiation exposure.
Device: Magnetic resonance imaging

SUMMARY:
Currently catheters used in heart catheterization procedures are guided throughout the heart chambers and blood vessels by pictures taken by x-rays. This technology exposes patients to radiation. With this study protocol the investigators will use MRI technology to take real-time pictures to navigate catheters throughout heart chambers. MRI uses electromagnetic energy; therefore, it does not expose participants to radiation energy.

DETAILED DESCRIPTION:
Participants undergo general anesthesia, and vascular access is obtained in the x-ray catheterization lab. Next the participant is transferred into the MRI scanner where a focused MRI examination is performed. Catheters are then guided into the heart chambers using real-time MRI guidance to perform conventional cardiac catheterization steps. If time allows, additional research MRI is performed before the participant is returned to the x-ray catheterization lab. If any MRI guided catheterization steps are unsuccessful, the clinically indicated step is performed after the participant returns to the x-ray catheterization lab using conventional x-ray guided pictures.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a medically necessary cardiovascular catheterization

Exclusion Criteria:

* Cardiovascular instability including hemodynamic instability (such as requiring significant vasoactive infusion support) or mechanical hemodynamic support.
* Women who are pregnant
* Women who are nursing and who do not plan to discard breast milk for 24 hours
* Patients with a contraindication to MRI scanning will be excluded. These contraindications include patients with the following devices:

  1. Central nervous system aneurysm clips
  2. Implanted neural stimulator
  3. Implanted cardiac pacemaker or defibrillator which are not MR safe or MR conditional according to the manufacturer
  4. Cochlear implant
  5. Ocular foreign body (e.g. metal shavings)
  6. Implanted Insulin pump
  7. Metal shrapnel or bullet

Exclusion criteria for Gadolinium (contrast agent)

1. Renal disease with estimated glomerular filtration rate < 30 ml/min/1.73 m2 body surface area

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Test the feasibility of navigating catheters into right heart structures using real-time MRI | At the end of each catheterization procedure through study completion,up to 5 years.
  Heart catheterization usually uses X-ray guidance. Using commercially available MRI-compatible catheters, the right heart catheterization procedure will be done using real-time magnetic resonance imaging (MRI). MRI guidance does not use X-ray radiation.

SECONDARY OUTCOMES:
Number of participants whose MRI cardiac catheterization procedure was prematurely terminated | At the end of each catheterization procedure through study completion,up to 5 years
  Premature termination will occur under the following circumstances:
  * Hemodynamic or other clinical instability
  * Technical failure of catheter procedure such as being unable to navigate the catheters to the heart chamber
  * Equipment malfunction
  * Any other circumstance that in the opinion of the Principal Investigator poses hazard to the research subject
Measurement of radiation exposure | End of study, 5 years.
  Comparison of radiation exposure in this cohort of subjects to historical controls undergoing matched invasive cardiology procedure at CNMC.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Kanter, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saikus CE, Lederman RJ. Interventional cardiovascular magnetic resonance imaging: a new opportunity for image-guided interventions. JACC Cardiovasc Imaging. 2009 Nov;2(11):1321-31. doi: 10.1016/j.jcmg.2009.09.002. PMID 19909937
- [Background] Ratnayaka K, Faranesh AZ, Guttman MA, Kocaturk O, Saikus CE, Lederman RJ. Interventional cardiovascular magnetic resonance: still tantalizing. J Cardiovasc Magn Reson. 2008 Dec 29;10(1):62. doi: 10.1186/1532-429X-10-62. PMID 19114017
- [Background] Guttman MA, Lederman RJ, Sorger JM, McVeigh ER. Real-time volume rendered MRI for interventional guidance. J Cardiovasc Magn Reson. 2002;4(4):431-42. doi: 10.1081/jcmr-120016382. PMID 12549231
- [Background] Guttman MA, Kellman P, Dick AJ, Lederman RJ, McVeigh ER. Real-time accelerated interactive MRI with adaptive TSENSE and UNFOLD. Magn Reson Med. 2003 Aug;50(2):315-21. doi: 10.1002/mrm.10504. PMID 12876708
- [Background] Peters DC, Lederman RJ, Dick AJ, Raman VK, Guttman MA, Derbyshire JA, McVeigh ER. Undersampled projection reconstruction for active catheter imaging with adaptable temporal resolution and catheter-only views. Magn Reson Med. 2003 Feb;49(2):216-22. doi: 10.1002/mrm.10390. PMID 12541240
- [Background] Guttman MA, Dick AJ, Raman VK, Arai AE, Lederman RJ, McVeigh ER. Imaging of myocardial infarction for diagnosis and intervention using real-time interactive MRI without ECG-gating or breath-holding. Magn Reson Med. 2004 Aug;52(2):354-61. doi: 10.1002/mrm.20174. PMID 15282818
- [Background] Peters DC, Guttman MA, Dick AJ, Raman VK, Lederman RJ, McVeigh ER. Reduced field of view and undersampled PR combined for interventional imaging of a fully dynamic field of view. Magn Reson Med. 2004 Apr;51(4):761-7. doi: 10.1002/mrm.20037. PMID 15065249
- [Background] de Silva R, Gutierrez LF, Raval AN, McVeigh ER, Ozturk C, Lederman RJ. X-ray fused with magnetic resonance imaging (XFM) to target endomyocardial injections: validation in a swine model of myocardial infarction. Circulation. 2006 Nov 28;114(22):2342-50. doi: 10.1161/CIRCULATIONAHA.105.598524. Epub 2006 Nov 13. PMID 17101858
- [Background] Guttman MA, Ozturk C, Raval AN, Raman VK, Dick AJ, DeSilva R, Karmarkar P, Lederman RJ, McVeigh ER. Interventional cardiovascular procedures guided by real-time MR imaging: an interactive interface using multiple slices, adaptive projection modes and live 3D renderings. J Magn Reson Imaging. 2007 Dec;26(6):1429-35. doi: 10.1002/jmri.21199. PMID 17968897
- [Background] Kocaturk O, Kim AH, Saikus CE, Guttman MA, Faranesh AZ, Ozturk C, Lederman RJ. Active two-channel 0.035'' guidewire for interventional cardiovascular MRI. J Magn Reson Imaging. 2009 Aug;30(2):461-5. doi: 10.1002/jmri.21844. PMID 19629968
- [Background] Kocaturk O, Saikus CE, Guttman MA, Faranesh AZ, Ratnayaka K, Ozturk C, McVeigh ER, Lederman RJ. Whole shaft visibility and mechanical performance for active MR catheters using copper-nitinol braided polymer tubes. J Cardiovasc Magn Reson. 2009 Aug 12;11(1):29. doi: 10.1186/1532-429X-11-29. PMID 19674464
- [Background] George AK, Derbyshire JA, Saybasili H, Saikus CE, Kocaturk O, Guttman MA, McVeigh ER, Lederman RJ, Faranesh AZ. Visualization of active devices and automatic slice repositioning ("SnapTo") for MRI-guided interventions. Magn Reson Med. 2010 Apr;63(4):1070-9. doi: 10.1002/mrm.22307. PMID 20373408
- [Background] Saybasili H, Derbyshire JA, Kellman P, Griswold MA, Ozturk C, Lederman RJ, Seiberlich N. RT-GROG: parallelized self-calibrating GROG for real-time MRI. Magn Reson Med. 2010 Jul;64(1):306-12. doi: 10.1002/mrm.22351. PMID 20577983
- [Background] Derbyshire JA, Herzka DA, McVeigh ER, Lederman RJ. Efficient implementation of hardware-optimized gradient sequences for real-time imaging. Magn Reson Med. 2010 Dec;64(6):1814-20. doi: 10.1002/mrm.22211. PMID 20878764
- [Background] Sampath S, Raval AN, Lederman RJ, McVeigh ER. High-resolution 3D arteriography of chronic total peripheral occlusions using a T1-W turbo spin-echo sequence with inner-volume imaging. Magn Reson Med. 2007 Jan;57(1):40-9. doi: 10.1002/mrm.21098. PMID 17152076
- [Background] Guttman MA, Raval AN, Lederman RJ, McVeigh ER. Real-time catheter-directed MRA with effective background suppression and persistent rendering. J Magn Reson Imaging. 2008 Aug;28(2):538-42. doi: 10.1002/jmri.21409. PMID 18666149
- [Background] Lederman RJ, Guttman MA, Peters DC, Thompson RB, Sorger JM, Dick AJ, Raman VK, McVeigh ER. Catheter-based endomyocardial injection with real-time magnetic resonance imaging. Circulation. 2002 Mar 19;105(11):1282-4. doi: 10.1161/01.cir.0000012425.71261.fc. PMID 11901036
- [Background] Dick AJ, Guttman MA, Raman VK, Peters DC, Pessanha BS, Hill JM, Smith S, Scott G, McVeigh ER, Lederman RJ. Magnetic resonance fluoroscopy allows targeted delivery of mesenchymal stem cells to infarct borders in Swine. Circulation. 2003 Dec 9;108(23):2899-904. doi: 10.1161/01.CIR.0000095790.28368.F9. Epub 2003 Dec 1. PMID 14656911
- [Background] Arepally A, Karmarkar PV, Weiss C, Rodriguez ER, Lederman RJ, Atalar E. Magnetic resonance image-guided trans-septal puncture in a swine heart. J Magn Reson Imaging. 2005 Apr;21(4):463-7. doi: 10.1002/jmri.20262. PMID 15779027
- [Background] Raman VK, Karmarkar PV, Guttman MA, Dick AJ, Peters DC, Ozturk C, Pessanha BS, Thompson RB, Raval AN, DeSilva R, Aviles RJ, Atalar E, McVeigh ER, Lederman RJ. Real-time magnetic resonance-guided endovascular repair of experimental abdominal aortic aneurysm in swine. J Am Coll Cardiol. 2005 Jun 21;45(12):2069-77. doi: 10.1016/j.jacc.2005.03.029. PMID 15963411
- [Background] Raval AN, Telep JD, Guttman MA, Ozturk C, Jones M, Thompson RB, Wright VJ, Schenke WH, DeSilva R, Aviles RJ, Raman VK, Slack MC, Lederman RJ. Real-time magnetic resonance imaging-guided stenting of aortic coarctation with commercially available catheter devices in Swine. Circulation. 2005 Aug 2;112(5):699-706. doi: 10.1161/CIRCULATIONAHA.105.542647. Epub 2005 Jul 25. PMID 16043639
- [Background] Raval AN, Karmarkar PV, Guttman MA, Ozturk C, Sampath S, DeSilva R, Aviles RJ, Xu M, Wright VJ, Schenke WH, Kocaturk O, Dick AJ, Raman VK, Atalar E, McVeigh ER, Lederman RJ. Real-time magnetic resonance imaging-guided endovascular recanalization of chronic total arterial occlusion in a swine model. Circulation. 2006 Feb 28;113(8):1101-7. doi: 10.1161/CIRCULATIONAHA.105.586727. Epub 2006 Feb 20. PMID 16490819
- [Background] Raval AN, Karmarkar PV, Guttman MA, Ozturk C, Desilva R, Aviles RJ, Wright VJ, Schenke WH, Atalar E, McVeigh ER, Lederman RJ. Real-time MRI guided atrial septal puncture and balloon septostomy in swine. Catheter Cardiovasc Interv. 2006 Apr;67(4):637-43. doi: 10.1002/ccd.20579. PMID 16532499
- [Background] Elagha AA, Kocaturk O, Guttman MA, Ozturk C, Kim AH, Burton GW, Kim JH, Raman VK, Raval AN, Wright VJ, Schenke WH, McVeigh ER, Lederman RJ. Real-time MR imaging-guided laser atrial septal puncture in swine. J Vasc Interv Radiol. 2008 Sep;19(9):1347-53. doi: 10.1016/j.jvir.2008.05.007. Epub 2008 Jul 21. PMID 18725098
- [Background] Dick AJ, Raman VK, Raval AN, Guttman MA, Thompson RB, Ozturk C, Peters DC, Stine AM, Wright VJ, Schenke WH, Lederman RJ. Invasive human magnetic resonance imaging: feasibility during revascularization in a combined XMR suite. Catheter Cardiovasc Interv. 2005 Mar;64(3):265-74. doi: 10.1002/ccd.20302. PMID 15736247
- [Background] Ratnayaka K, Faranesh AZ, Hansen MS, Stine AM, Halabi M, Barbash IM, Schenke WH, Wright VJ, Grant LP, Kellman P, Kocaturk O, Lederman RJ. Real-time MRI-guided right heart catheterization in adults using passive catheters. Eur Heart J. 2013 Feb;34(5):380-9. doi: 10.1093/eurheartj/ehs189. Epub 2012 Aug 1. PMID 22855740
- [Background] Kleinerman RA. Cancer risks following diagnostic and therapeutic radiation exposure in children. Pediatr Radiol. 2006 Sep;36 Suppl 2(Suppl 2):121-5. doi: 10.1007/s00247-006-0191-5. PMID 16862418
- [Background] Andreassi MG, Ait-Ali L, Botto N, Manfredi S, Mottola G, Picano E. Cardiac catheterization and long-term chromosomal damage in children with congenital heart disease. Eur Heart J. 2006 Nov;27(22):2703-8. doi: 10.1093/eurheartj/ehl014. Epub 2006 May 22. PMID 16717079
- [Background] Niendorf HP, Dinger JC, Haustein J, Cornelius I, Alhassan A, Clauss W. Tolerance data of Gd-DTPA: a review. Eur J Radiol. 1991 Jul-Aug;13(1):15-20. doi: 10.1016/0720-048x(91)90049-2. PMID 1889423
- [Background] Niendorf HP, Haustein J, Cornelius I, Alhassan A, Clauss W. Safety of gadolinium-DTPA: extended clinical experience. Magn Reson Med. 1991 Dec;22(2):222-8; discussion 229-32. doi: 10.1002/mrm.1910220212. PMID 1812350
- [Background] Niendorf HP, Haustein J, Louton T, Beck W, Laniado M. Safety and tolerance after intravenous administration of 0.3 mmol/kg Gd-DTPA. Results of a randomized, controlled clinical trial. Invest Radiol. 1991 Nov;26 Suppl 1:S221-3; discussion S232-5. doi: 10.1097/00004424-199111001-00075. No abstract available. PMID 1808134
- [Background] Kiringoda R, Thurm AE, Hirschtritt ME, Koziol D, Wesley R, Swedo SE, O'Grady NP, Quezado ZM. Risks of propofol sedation/anesthesia for imaging studies in pediatric research: eight years of experience in a clinical research center. Arch Pediatr Adolesc Med. 2010 Jun;164(6):554-60. doi: 10.1001/archpediatrics.2010.75. PMID 20530306
- [Background] Schwartz GJ, Haycock GB, Edelmann CM Jr, Spitzer A. A simple estimate of glomerular filtration rate in children derived from body length and plasma creatinine. Pediatrics. 1976 Aug;58(2):259-63. PMID 951142
- [Background] Beels L, Bacher K, De Wolf D, Werbrouck J, Thierens H. gamma-H2AX foci as a biomarker for patient X-ray exposure in pediatric cardiac catheterization: are we underestimating radiation risks? Circulation. 2009 Nov 10;120(19):1903-9. doi: 10.1161/CIRCULATIONAHA.109.880385. Epub 2009 Oct 26. PMID 19858412
- [Background] Haustein J, Laniado M, Niendorf HP, Louton T, Beck W, Planitzer J, Schoffel M, Reiser M, Kaiser W, Schorner W, et al. Triple-dose versus standard-dose gadopentetate dimeglumine: a randomized study in 199 patients. Radiology. 1993 Mar;186(3):855-60. doi: 10.1148/radiology.186.3.8430199.
- [Background] Niendorf HP, Alhassan A, Geens VR, Clauss W. Safety review of gadopentetate dimeglumine. Extended clinical experience after more than five million applications. Invest Radiol. 1994 Jun;29 Suppl 2:S179-82. doi: 10.1097/00004424-199406001-00059. No abstract available. PMID 7928222
- [Background] Dillman JR, Ellis JH, Cohan RH, Strouse PJ, Jan SC. Frequency and severity of acute allergic-like reactions to gadolinium-containing i.v. contrast media in children and adults. AJR Am J Roentgenol. 2007 Dec;189(6):1533-8. doi: 10.2214/AJR.07.2554. PMID 18029897
- [Background] Sundgren PC, Leander P. Is administration of gadolinium-based contrast media to pregnant women and small children justified? J Magn Reson Imaging. 2011 Oct;34(4):750-7. doi: 10.1002/jmri.22413. PMID 21928308
- [Background] Deo A, Fogel M, Cowper SE. Nephrogenic systemic fibrosis: a population study examining the relationship of disease development to gadolinium exposure. Clin J Am Soc Nephrol. 2007 Mar;2(2):264-7. doi: 10.2215/CJN.03921106. Epub 2007 Feb 7. PMID 17699423
- [Background] Tello R, Mitchell PJ, Melhem ER, Witte D, Thomson KR. Interventional catheter magnetic resonance angiography with a conventional 1.5-T magnet: work in progress. Australas Radiol. 1999 Nov;43(4):435-9. doi: 10.1046/j.1440-1673.1999.00706.x. PMID 10901954
- [Background] Paetzel C, Zorger N, Seitz J, Volk M, Nitz WR, Herold T, Feuerbach S, Lenhart M. Intraarterial contrast material-enhanced magnetic resonance angiography of the aortoiliac system. J Vasc Interv Radiol. 2004 Sep;15(9):981-4. doi: 10.1097/01.RVI.0000133700.86048.3D. PMID 15361566
- [Background] Paetzel C, Zorger N, Volk M, Herold T, Seitz J, Nitz WR, Feuerbach S, Hamer O, Lenhart M. Intra-arterial magnetic resonance angiography of the iliac arteries: clinical experience using two different protocols. Acta Radiol. 2005 May;46(3):250-5. doi: 10.1080/02841850510021030. PMID 15981721
- [Background] Schulte AC, Bongartz G, Huegli R, Aschwanden M, Jaeger KA, Ostheim-Dzerowycz W, Jacob AL, Bilecen D. Intraarterial versus IV gadolinium injections for MR angiography: quantitative and qualitative assessment of the infrainguinal arteries. AJR Am J Roentgenol. 2005 Sep;185(3):735-40. doi: 10.2214/ajr.185.3.01850735. PMID 16120927
- [Background] Bozlar U, Norton PT, Turba UC, Hagspiel KD. Novel technique for evaluating complex pelvic arteriovenous malformations with catheter-directed subtracted MR angiography. J Vasc Interv Radiol. 2007 Jul;18(7):920-3. doi: 10.1016/j.jvir.2007.04.003. PMID 17609455
- [Background] Schmitt B, Steendijk P, Lunze K, Ovroutski S, Falkenberg J, Rahmanzadeh P, Maarouf N, Ewert P, Berger F, Kuehne T. Integrated assessment of diastolic and systolic ventricular function using diagnostic cardiac magnetic resonance catheterization: validation in pigs and application in a clinical pilot study. JACC Cardiovasc Imaging. 2009 Nov;2(11):1271-81. doi: 10.1016/j.jcmg.2009.09.007. PMID 19909930
- [Background] Larose E, Yeghiazarians Y, Libby P, Yucel EK, Aikawa M, Kacher DF, Aikawa E, Kinlay S, Schoen FJ, Selwyn AP, Ganz P. Characterization of human atherosclerotic plaques by intravascular magnetic resonance imaging. Circulation. 2005 Oct 11;112(15):2324-31. doi: 10.1161/CIRCULATIONAHA.105.538942. Epub 2005 Oct 3. PMID 16203910
- [Background] Razavi R, Hill DL, Keevil SF, Miquel ME, Muthurangu V, Hegde S, Rhode K, Barnett M, van Vaals J, Hawkes DJ, Baker E. Cardiac catheterisation guided by MRI in children and adults with congenital heart disease. Lancet. 2003 Dec 6;362(9399):1877-82. doi: 10.1016/S0140-6736(03)14956-2. PMID 14667742
- [Background] Miquel ME, Hegde S, Muthurangu V, Corcoran BJ, Keevil SF, Hill DL, Razavi RS. Visualization and tracking of an inflatable balloon catheter using SSFP in a flow phantom and in the heart and great vessels of patients. Magn Reson Med. 2004 May;51(5):988-95. doi: 10.1002/mrm.20041. PMID 15122681
- [Background] Muthurangu V, Taylor A, Andriantsimiavona R, Hegde S, Miquel ME, Tulloh R, Baker E, Hill DL, Razavi RS. Novel method of quantifying pulmonary vascular resistance by use of simultaneous invasive pressure monitoring and phase-contrast magnetic resonance flow. Circulation. 2004 Aug 17;110(7):826-34. doi: 10.1161/01.CIR.0000138741.72946.84. Epub 2004 Aug 9. PMID 15302793
- [Background] Kuehne T, Yilmaz S, Steendijk P, Moore P, Groenink M, Saaed M, Weber O, Higgins CB, Ewert P, Fleck E, Nagel E, Schulze-Neick I, Lange P. Magnetic resonance imaging analysis of right ventricular pressure-volume loops: in vivo validation and clinical application in patients with pulmonary hypertension. Circulation. 2004 Oct 5;110(14):2010-6. doi: 10.1161/01.CIR.0000143138.02493.DD. Epub 2004 Sep 27. PMID 15451801
- [Background] Kuehne T, Yilmaz S, Schulze-Neick I, Wellnhofer E, Ewert P, Nagel E, Lange P. Magnetic resonance imaging guided catheterisation for assessment of pulmonary vascular resistance: in vivo validation and clinical application in patients with pulmonary hypertension. Heart. 2005 Aug;91(8):1064-9. doi: 10.1136/hrt.2004.038265. PMID 16020598
- [Background] Paetzel C, Zorger N, Bachthaler M, Hamer OW, Stehr A, Feuerbach S, Lenhart M, Volk M, Herold T, Kasprzak P, Nitz WR. Magnetic resonance-guided percutaneous angioplasty of femoral and popliteal artery stenoses using real-time imaging and intra-arterial contrast-enhanced magnetic resonance angiography. Invest Radiol. 2005 May;40(5):257-62. doi: 10.1097/01.rli.0000159876.09033.2e. PMID 15829822
- [Background] Kee ST, Ganguly A, Daniel BL, Wen Z, Butts K, Shimikawa A, Pelc NJ, Fahrig R, Dake MD. MR-guided transjugular intrahepatic portosystemic shunt creation with use of a hybrid radiography/MR system. J Vasc Interv Radiol. 2005 Feb;16(2 Pt 1):227-34. doi: 10.1097/01.RVI.0000143766.08029.6E. PMID 15713923
- [Background] Krueger JJ, Ewert P, Yilmaz S, Gelernter D, Peters B, Pietzner K, Bornstedt A, Schnackenburg B, Abdul-Khaliq H, Fleck E, Nagel E, Berger F, Kuehne T. Magnetic resonance imaging-guided balloon angioplasty of coarctation of the aorta: a pilot study. Circulation. 2006 Feb 28;113(8):1093-100. doi: 10.1161/CIRCULATIONAHA.105.578112. Epub 2006 Feb 20. PMID 16490822
- [Background] Muthurangu V, Atkinson D, Sermesant M, Miquel ME, Hegde S, Johnson R, Andriantsimiavona R, Taylor AM, Baker E, Tulloh R, Hill D, Razavi RS. Measurement of total pulmonary arterial compliance using invasive pressure monitoring and MR flow quantification during MR-guided cardiac catheterization. Am J Physiol Heart Circ Physiol. 2005 Sep;289(3):H1301-6. doi: 10.1152/ajpheart.00957.2004. Epub 2005 May 6. PMID 15879483
- [Background] Huegli RW, Aschwanden M, Kos S, Rasmus M, Jaeger K, Jacob AL, Bilecen D. Diagnostic pitfalls in postinterventional intraarterial magnetic resonance angiography after recanalization of femoropopliteal arterial occlusions. Acta Radiol. 2008 Dec;49(10):1129-36. doi: 10.1080/02841850802508942. PMID 19031180
- [Background] Tzifa A, Krombach GA, Kramer N, Kruger S, Schutte A, von Walter M, Schaeffter T, Qureshi S, Krasemann T, Rosenthal E, Schwartz CA, Varma G, Buhl A, Kohlmeier A, Bucker A, Gunther RW, Razavi R. Magnetic resonance-guided cardiac interventions using magnetic resonance-compatible devices: a preclinical study and first-in-man congenital interventions. Circ Cardiovasc Interv. 2010 Dec;3(6):585-92. doi: 10.1161/CIRCINTERVENTIONS.110.957209. Epub 2010 Nov 23. PMID 21098745
- [Background] Sommer P, Grothoff M, Eitel C, Gaspar T, Piorkowski C, Gutberlet M, Hindricks G. Feasibility of real-time magnetic resonance imaging-guided electrophysiology studies in humans. Europace. 2013 Jan;15(1):101-8. doi: 10.1093/europace/eus230. Epub 2012 Jul 31. PMID 22849974
- [Background] Nordbeck P, Beer M, Kostler H, Ladd ME, Quick HH, Bauer WR, Ritter O. Cardiac catheter ablation under real-time magnetic resonance guidance. Eur Heart J. 2012 Aug;33(15):1977. doi: 10.1093/eurheartj/ehs139. Epub 2012 Jun 7. No abstract available. PMID 22677138
- [Background] Nazarian S, Kolandaivelu A, Zviman MM, Meininger GR, Kato R, Susil RC, Roguin A, Dickfeld TL, Ashikaga H, Calkins H, Berger RD, Bluemke DA, Lardo AC, Halperin HR. Feasibility of real-time magnetic resonance imaging for catheter guidance in electrophysiology studies. Circulation. 2008 Jul 15;118(3):223-9. doi: 10.1161/CIRCULATIONAHA.107.742452. Epub 2008 Jun 23. PMID 18574048
- [Background] Manke C, Nitz WR, Djavidani B, Strotzer M, Lenhart M, Volk M, Feuerbach S, Link J. MR imaging-guided stent placement in iliac arterial stenoses: a feasibility study. Radiology. 2001 May;219(2):527-34. doi: 10.1148/radiology.219.2.r01ma03527. PMID 11323483
- [Background] Hofmann LV, Liddell RP, Eng J, Wasserman BA, Arepally A, Lee DS, Bluemke DA. Human peripheral arteries: feasibility of transvenous intravascular MR imaging of the arterial wall. Radiology. 2005 May;235(2):617-22. doi: 10.1148/radiol.2352040340. PMID 15858101
- [Background] Araki T, Aoki S, Ishigame K, Kumagai H, Nanbu A, Hori M, Ueki J, Komiyama T, Araki T. MR-guided intravascular catheter manipulation: feasibility of both active and passive tracking in experimental study and initial clinical applications. Radiat Med. 2002 Jan-Feb;20(1):1-8. PMID 12002598
- [Derived] Ratnayaka K, Kanter JP, Faranesh AZ, Grant EK, Olivieri LJ, Cross RR, Cronin IF, Hamann KS, Campbell-Washburn AE, O'Brien KJ, Rogers T, Hansen MS, Lederman RJ. Radiation-free CMR diagnostic heart catheterization in children. J Cardiovasc Magn Reson. 2017 Sep 6;19(1):65. doi: 10.1186/s12968-017-0374-2. PMID 28874164